CLINICAL TRIAL: NCT05685459
Title: Position and Communication Skills Simulation: Comparison of Two Simulation Models in Nursing Student
Brief Title: Position and Communication Skills Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, özlem doğu, Associate Professor, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Comparison Simulation Models
Record Dates: First submitted 2022-12-24; First posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Comparing to Effect Two Simulation Models
Keywords: Standardized patient; Simulation; Nurse; Positioning skills; Communication skills

STUDY DESIGN:
Intervention Model Description: The population of the study consisted of 112 second-semester nursing students who took the "Nursing Fundamentals" course in the spring semester of the 2021-2022 academic year, and the sample included volunteers who took the course for the first time. A power analysis was performed on the G*Power (v3.1.7) software to determine the sample size. The power of a study is expressed as 1-β (β = probability of type II error), and in general, studies should have 80% power. According to Cohen's effect size coefficients, assuming that the evaluations between two independent groups would have a large effect size (d = 0.8), the sample size was calculated as 60 subjects. Students were randomly assigned to groups using computer software.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The students involved in the intervention group were divided into subgroups, and the simulation was carried out using standardized patients. Each subgroup consisted of two students. Students were asked to practice supine and lateral recumbent positions in each scenario.
  Interventions: Other: Standard patient simulation model
- Control (No Intervention): The students in the control group were divided into subgroups and practised the supine position and the lateral recumbent position with a high-fidelity manikin. Each subgroup consisted of two students. The applications lasted 5-10 minutes for each group, and after the applications, the debriefing phase was conducted, which lasted 20 minutes.

INTERVENTIONS:
Other: Standard patient simulation model — Nursing students were trained with a standard patient simulation model for position and communication skills education.
  Arms: Intervention

SUMMARY:
The goal of this study was to compare two different simulation applications in developing the positioning skill, one of the most common nursing practices, and the communication skill, which forms the basis of nursing practices.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* First-year nursing students
* Not have training in simulation

Exclusion Criteria:

* Not meeting the inclusion criteria

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Comparing of two simulation models | 1 month
  Describing the performance scores of the students in the standardized patient group and the high-fidelity simulation manikin group.
  The checklist consisted of 20 steps. The student scored "0" if "the step was not applied at all" or "the step was applied incorrectly." If the "step was not fully implemented", it was graded with "1" point, and "if the step was performed correctly and completely," it was graded with "2" points. Checklists were filled out by an independent observer, who was not a researcher. Scores that can be obtained from the skill checklist ranged between 0 and 80, which were converted to 100 points.

SECONDARY OUTCOMES:
Therapeutic Communication Skills Questionnaire for Nursing Students | 1 month
  Therapeutic Communication Skills Questionnaire for Nursing Students: It is a 7-point Likert-type scale and consists of 16 items and three sub-dimensions. The highest total score that can be obtained from the scale is 112, which shows high therapeutic communication skills.
The Student Satisfaction and Self-Confidence Scale | 1 month
  The Student Satisfaction and Self-Confidence Scale: The scale has a 5-point Likert-type evaluation structure and consists of 13 items and two sub-dimensions. The highest total score that can be obtained from the scale is 65, which means high satisfaction and self-confidence.

CONTACTS AND LOCATIONS:
Overall Officials: Şengül ÜZEN CURA, Doctorate, Study Chair — Çanakkale On Sekiz Mart University
Locations (1):
- Ozlem Dogu, Sakarya, Serdivan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berman, A.,Snyder, S., &Frandsen, G. (2016). Fundamentals of nursing: concept, process, andpractice (10th ed.). New Jersey: Pearson.
- [Background] Potter, P.A., Perry, A.G., &Stockert, P.A. Fundamentals of nursing(10, revised ed.). (2021). St. Louis:Elsevier.
- [Result] Wilfong DN, Falsetti DJ, McKinnon JL, Daniel LH, Wan QC. The effects of virtual intravenous and patient simulator training compared to the traditional approach of teaching nurses: a research project on peripheral i.v. catheter insertion. J Infus Nurs. 2011 Jan-Feb;34(1):55-62. doi: 10.1097/NAN.0b013e31820219e2. PMID 21239952
- [Result] McWilliams LA, Malecha A. Comparing Intravenous Insertion Instructional Methods with Haptic Simulators. Nurs Res Pract. 2017;2017:4685157. doi: 10.1155/2017/4685157. Epub 2017 Jan 29. PMID 28250987
- [Result] Vidal VL, Ohaeri BM, John P, Helen D. Virtual reality and the traditional method for phlebotomy training among college of nursing students in Kuwait: implications for nursing education and practice. J Infus Nurs. 2013 Sep-Oct;36(5):349-55. doi: 10.1097/NAN.0b013e318243172f. PMID 24006114
- [Result] Ignacio J, Dolmans D, Scherpbier A, Rethans JJ, Chan S, Liaw SY. Comparison of standardized patients with high-fidelity simulators for managing stress and improving performance in clinical deterioration: A mixed methods study. Nurse Educ Today. 2015 Dec;35(12):1161-8. doi: 10.1016/j.nedt.2015.05.009. Epub 2015 May 23. PMID 26047602
- [Result] Uzen Cura S, Kocatepe V, Yildirim D, Kucukakgun H, Atay S, Unver V. Examining Knowledge, Skill, Stress, Satisfaction, and Self-Confidence Levels of Nursing Students in Three Different Simulation Modalities. Asian Nurs Res (Korean Soc Nurs Sci). 2020 Aug;14(3):158-164. doi: 10.1016/j.anr.2020.07.001. Epub 2020 Jul 9. PMID 32653666
- [Result] Doolen J, Giddings M, Johnson M, Guizado de Nathan G, O Badia L. An evaluation of mental health simulation with standardized patients. Int J Nurs Educ Scholarsh. 2014 Mar 12;11:/j/ijnes.2014.11.issue-1/ijnes-2013-0075/ijnes-2013-0075.xml. doi: 10.1515/ijnes-2013-0075. PMID 24620017
- [Result] Quail M, Brundage SB, Spitalnick J, Allen PJ, Beilby J. Student self-reported communication skills, knowledge and confidence across standardised patient, virtual and traditional clinical learning environments. BMC Med Educ. 2016 Feb 27;16:73. doi: 10.1186/s12909-016-0577-5. PMID 26919838
- [Result] Olaussen C, Heggdal K, Tvedt CR. Elements in scenario-based simulation associated with nursing students' self-confidence and satisfaction: A cross-sectional study. Nurs Open. 2019 Sep 27;7(1):170-179. doi: 10.1002/nop2.375. eCollection 2020 Jan. PMID 31871700
- [Result] MacLean S, Kelly M, Geddes F, Della P. Use of simulated patients to develop communication skills in nursing education: An integrative review. Nurse Educ Today. 2017 Jan;48:90-98. doi: 10.1016/j.nedt.2016.09.018. Epub 2016 Sep 28. PMID 27741440
- [Result] Cabanero-Martinez MJ, Garcia-Sanjuan S, Escribano S, Fernandez-Alcantara M, Martinez-Riera JR, Julia-Sanchis R. Mixed-method study on the satisfaction of a high-fidelity simulation program in a sample of nursing-degree students. Nurse Educ Today. 2021 May;100:104858. doi: 10.1016/j.nedt.2021.104858. Epub 2021 Mar 6. PMID 33713986
- See also: A Technological Step in Nursing Education: Intramuscular Injection ventro-sim — https://jag.journalagent.com/jaren/pdfs/JAREN_2_2_103_108.pdf
- See also: Using standardized patients to improve the hygiene care skills of first-year nursing students: A randomized controlled trial — https://doi.org/10.1016/j.colegn.2018.03.005
- See also: Effects of Simulation-based Education on Communication Skill and Clinical Competence in Maternity Nursing Practicum — https://koreascience.kr/article/JAKO201207339091888.pdf